CLINICAL TRIAL: NCT00879294
Title: The Effect of Gum Chewing on Postoperative Ileus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CR1_IRB00005677
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-07

CONDITIONS: Perforated Appendicitis
Keywords: Perforated appendicitis; Ruptured appendicitis; Acute appendicitis with perforation
MeSH Terms: conditions — Appendicitis | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- 1 Wristband (Sham Comparator): Some patients will be randomized to wear a motion sickness wristband which does not have any drug effect.
  Interventions: Device: Motion sickness wristband
- Chewing Gum (Experimental): Patients will be randomized to use chewing gum after surgery.
  Interventions: Dietary Supplement: Chewing Gum
- Control (No Intervention): Usual post-operative care.

INTERVENTIONS:
Device: Motion sickness wristband — No drugs are involved.
  Arms: 1 Wristband
Dietary Supplement: Chewing Gum — Patients will be asked to chew gum for 20 minutes, four times daily.
  Arms: Chewing Gum

SUMMARY:
The purpose of this study is to see if chewing gum after surgery for perforated appendicitis will shorten the time of intestinal dysfunction.

DETAILED DESCRIPTION:
After operations for a ruptured appendix, children are usually not allowed to eat or drink anything. This is because the infection inside the abdomen and the manipulation of the intestines during the operation cause the bowels to stop their normal movement. The resulting lack of bowel function is called an "ileus". When this occurs, intestinal secretions and anything taken in by mouth can become backed up, causing bloating, abdominal pain, nausea and vomiting. Children are not allowed to eat or drink anything during this time and require fluid hydration through an IV or even nutrition through an IV. This ileus usually lasts an average of 4-5 days, and can sometimes delay the discharge of children who are otherwise ready to go. The purpose of this research study is to determine if simple things, like gum chewing or anti-motion sickness bracelets can help speed the time it takes for the bowels to begin working after an operation for a ruptured appendix. Because the gum is not swallowed, it does not have the same effects as eating and drinking would on someone with an ileus. The same is true for the anti-motion sickness bracelets. Yet, it is thought that the chewing action from gum may stimulate the intestines into thinking that food is on the way and cause them to start working sooner than they otherwise might. The same may be true for the bracelets, and some studies show them to be helpful with nausea after surgery. Nevertheless, the effects of a bracelet on postoperative ileus are unproven.

ELIGIBILITY:
Inclusion Criteria:

* any child who has undergone appendectomy for perforated appendicitis

Exclusion Criteria:

* age less than or equal to 5 years
* unable to chew gum safely
* interval appendectomy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Time to resolution of post-operative ileus. | 1-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pranikoff, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Brenner Children's Hospital, Winston-Salem, North Carolina, United States